CLINICAL TRIAL: NCT06907446
Title: Comparison of BARD Max Core 18g Needle With Uro1 SUREcore 18g Needle in Targeted Prostate Biopsies
Brief Title: Comparison of New SUREcore Biopsy of Needle to Standard of Care During Transperineal Prostate Biopsies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2262703
Record Dates: First submitted 2025-03-10; First posted 2025-04-02 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single arm study comparing two different needle biopsy systems for prostate biopsy (Other)
  Interventions: Diagnostic Test: Comparison of Biopsy Needle Types for Prostate Biopsy

INTERVENTIONS:
Diagnostic Test: Comparison of Biopsy Needle Types for Prostate Biopsy — Each patient will undergo a standard of care prostate biopsy according to the clinical indication alternating between the SureCore and standard Bard needle

SUMMARY:
To study a novel biopsy needle system for performing transperineal prostate biopsy. Prostate biopsy remains the standard approach for prostate cancer detection. While pre-biopsy MRI allows for targeting of visible lesions, systemic or 'off target' samples are recommended due to the well-recognized risk of undegrading and under sampling with current commercially available needles. The SureCore plus single-use biopsy needle produces a more intact tissue core with a same caliber 18g needle with ~21% more tissue per core in pre-clinical studies. This research study will determine if a new biopsy needle designed to produce more robust tissue cores per sample can improve detection and characterization of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than age of 18 undergoing prostate biopsy

Exclusion Criteria:

* Unable to consent
* Any comorbidity that, in the opinion of the investigator, could compromise protocol objectives
* Prisoners

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients diagnosed with prostate cancer and histological grade of cancer detected | From prostate biopsy procedure through study completion up to 1 year
  The primary outcome will evaluate whether cancer is detected on final pathological analysis. This will include the grade of cancer, percentage of core involved, and compare between the two needles.

SECONDARY OUTCOMES:
Quality of Biopsy Specimen Obtained at Time of Prostate Biopsy | From prostate biopsy procedure through study completion up to 1 year
  The secondary outcomes will look at the quality of specimen including fragmentation, tortuosity, and spatial orientation of the sample.
Length of time necessary to diagnose the tissue sample | Diagnosis within 10 days of the biopsy
  Time required from collection of specimen to final diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Departments of Urologic Oncology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No